CLINICAL TRIAL: NCT00413296
Title: A Double-Blind Discontinuation Study of Levetiracetam in Post- Traumatic Stress Disorder
Brief Title: Levetiracetam in Post-Traumatic Stress Disorder
Acronym: PTSD
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: UCB Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pro00007843; 7031-05-4R0 (Other: DUMC)
Record Dates: First submitted 2006-12-18; First posted 2006-12-19 (Estimated); Last update posted 2014-07-21 (Estimated); Status verified 2010-06

CONDITIONS: Post-Traumatic Stress Disorder
Keywords: PTSD; Anxiety; Pharmacotherapy; Levetiracetam; Relapse prevention
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Anxiety Disorders | interventions — Levetiracetam

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Placebo Comparator): Tablets, no active ingredient, 1-6 tablets/day for 12 wks in the 2 nd phase of the trial.
  Interventions: Drug: Placebo
- 2 (Active Comparator): Levetiracetam, 500mg (1-6 tablets /day) for 12 wks in the 2nd phase of the study.
  Interventions: Drug: levetiracetam; Drug: Levetriracetam

INTERVENTIONS:
Drug: levetiracetam — Tablets, dosage 500 mg each ( 1-6 tablets/day)for20 wks
  Other Names: Keppra
  Arms: 2
Drug: Placebo — Placebo, Tablets, no active ingredient in the tablets, (1-6tablets/day)for 12 wks in the 2nd phase of the study.
  Arms: 1
Drug: Levetriracetam — Tablets, 500 mg each (1-6 tablets/day) for 8 wks during the open label phase and for 12 wks during the 2nd phase of the study.
  Other Names: Keppra
  Arms: 2

SUMMARY:
The purpose of this study is to evaluate the short-term efficacy and safety of levetiracetam in post-traumatic stress disorder (PTSD) and to evaluate continuation effects of levetiracetam in preventing PTSD relapse. The hypothesis is that levetiracetam will be safe and effective in preventing relapse of PTSD.

DETAILED DESCRIPTION:
This is an investigator-initiated, single site study, consisting of two phases: 8 weeks of open label treatment with levetiracetam (500-2000 mg/day) in patients with PTSD, and in those who demonstrate at least minimal improvement, 12 weeks of randomized, double-blind treatment with either levetiracetam or matching placebo.

ELIGIBILITY:
Inclusion Criteria:

* ages 18-65
* primary diagnosis of PTSD based on DSM-IV criteria and assessed by the MINI International Neuropsychiatric Interview (MINI)
* Davidson Trauma Scale (DTS) score of at least 40 on screening
* ability to provide written informed consent

Exclusion Criteria:

* any primary DSM-IV Axis I disorder other than PTSD
* substance abuse during the last 6 months
* a clinically unstable medical condition or clinically significant laboratory abnormalities
* suicide risk or serious suicide attempt during the last year
* concurrent use of psychotropic medications including benzodiazepines, barbiturates, antiepileptic drugs, antidepressants, buspirone, dietary supplements or herbal or homeopathic remedies with psychotropic effects
* recent (within the last 3 months) initiation of cognitive behavioral therapy
* failure of a previous trial of levetiracetam at 2000 mg/day
* pregnancy or lactation
* women of childbearing potential who are unwilling to practice an acceptable method of contraception

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2005-11; Primary Completion 2007-09 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Clinical Global Impressions - Improvement (CGI-I) | 20 wks

SECONDARY OUTCOMES:
Davidson Trauma Scale (DTS) | 20 wks
Hospital Anxiety and Depression Scale (HADS) | 20 wks
Connor-Davidson Resilience Scale (CD-RISC) | 20 wks
36-item Short Form Health Survey (SF-36) | 20 wks
Pittsburgh Sleep Quality Index | 20 wks
Work Productivity and Activity Improvement Questionnaire (WPAI) | 20 wks
Sheehan Disability Inventory (SDI) | 20 wks

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Davidson, M.D., Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States